CLINICAL TRIAL: NCT07197151
Title: CYFIP1 and PKM2 Synergistically Regulate ROS and Glycolysis in Colorectal Cancer Through the AKT/mTOR/HIF-1α Cascad
Status: Completed | Type: Observational
Sponsor: hui hou (Other)
Responsible Party: Sponsor-Investigator, hui hou, Chief Physician, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Other Study IDs: 280211; 2022zhyx-C39 (Other Grant/Funding Number: Translational Medicine Research of Anhui Province)
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer (CRC); Specimens Are to be Collected From Subjects Who Are Having or Have Had a Fluid or Tissue Removed, a Biopsy or a Blood or Bone Marrow Draw
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Colorectal cancer tissue specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Perform surgery on patients with colorectal cancer and collect cancer and adjacent tissue specimens — Perform surgery on patients with colorectal cancer and collect cancer and adjacent tissue specimens

SUMMARY:
Collect some tumor tissue specimens from patients who have undergone colorectal cancer surgery and conduct experiments such as immunohistochemistry to observe the expression of related genes in colorectal cancer.

DETAILED DESCRIPTION:
We need to collect postoperative specimens and adjacent normal tissue specimens from patients with colorectal cancer for immunohistochemical staining. There is no need to conduct any other grouping of the patients.

ELIGIBILITY:
Inclusion Criteria:(1) Patients diagnosed with colorectal cancer who received surgical treatment and postoperative chemotherapy (2) Patients who were conscious of their condition and voluntarily participated (3) No other serious underlying diseases

Exclusion Criteria:(1) Concurrent other serious chronic diseases or organ damage (2) Diagnosed with benign colorectal tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with colorectal cancer who have undergone surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Immunohistochemical determination of the expression levels of related genes | 2022.09-2025.09

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
The collected information includes the patient's personal details. It will still be needed for further experiments and cannot be shared for the time being.

DOCUMENTS (1):
  • Study Protocol (2025-09-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT07197151/Prot_000.pdf